CLINICAL TRIAL: NCT04094012
Title: Comparing Incidence Rate of Systemic Drug Reactions Under 3HP and 1HP Regimen for Latent Tuberculosis Infection Treatment: a Pragmatic Multicenter Randomized Control Trial
Brief Title: Risk of SDRs Under 3HP and 1HP Regimen for LTBI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201812127MINB
Record Dates: First submitted 2019-09-03; First posted 2019-09-18 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Latent Tuberculosis Infection
Keywords: isoniazid; latent tuberculosis infection; preventive therapy; rifapentine; systemic drug reaction; therapeutic drug monitoring
MeSH Terms: conditions — Latent Tuberculosis | interventions — Isoniazid; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-months weekly RPT plus INH (3HP) (Active Comparator): weekly RPT (900 mg for participants with body weight >50.0 kg; 750 mg for 32.1-50.0 kg; 600 mg for 25.1-32.0 kg; and 450 mg for 14.1-25.0 kg) plus INH (dose: 15 mg/kg, rounded up to nearest 150 mg; maximum 900 mg) for a total of 12 doses.
  Interventions: Drug: isoniazid and rifapentine
- 1-month daily RPT plus INH (1HP) (Experimental): daily RPT (dose: 600 mg for participants with body weight ≥45.0 kg; 450 mg for <45.0 kg) plus INH (dose: 300 mg) for a total of 28 days.
  Interventions: Drug: isoniazid and rifapentine

INTERVENTIONS:
Drug: isoniazid and rifapentine — This prospective multicenter randomized control trial (RCT) will be conducted on LTBI cases (see 2. Study population) to compare the risk of SDRs under conventional 3HP regimen (Arm 1: 3HP) and a new regimen consisting of daily RPT (10 mg/kg) plus INH (5 mg/kg) for 1 month (Arm 2: 1HP)
  Other Names: INH/RPT

SUMMARY:
Successful implement of preventive therapy for subjects with latent tuberculosis infection (LTBI) is the critical step for elimination of tuberculosis (TB). The major obstacle of traditional preventive therapy is the unacceptable long treatment duration, taking isoniazid 5mg/kg daily for a total of 9 months (9H), thus seriously compromising its acceptability. With the introduction of 12-doses weekly high-dose (15 mg/kg) rifapentine plus isoniazid (3HP regimen), the completion rate of 3HP has be shown to be much higher than 9H. However, 4.9% to 9.1% of LTBI cases who received 3HP failed to complete treatment because of side effects. Systemic drug reactions (SDRs), even hypotension and shock, under 3HP treatment are higher than 9H treatment.

A recent study in HIV patients demonstrated that a new short-term regimen, consisting of isoniazid 5mg/kg plus rifapentine 10mg/kg daily for one month (1HP), has a similar risk of adverse reactions as 3HP. Clinical study with head-to-head comparison between 3HP and 1HP, however, remains lacking.

The prospective multicenter study is conducted to investigate whether risk of SDRs under 1HP is lower than that under 3HP.

Hypothesis: 1HP has a lower incidence rate of SDRs than 3HP

Objectives:

1. To compare the risk of SDRs in 1HP treatment and in 3HP treatment
2. To explore side effect profile of 1HP

Methods:

This multicenter randomized control trial will compare the risk of SDRs under conventional 3HP regimen (Arm 1: 3HP), and a new regimen consisting of daily rifapentine (10 mg/kg) plus isoniazid (5 mg/kg) for 1 month (Arm 2: 1HP).

DETAILED DESCRIPTION:
Tuberculosis (TB) remains one of the deadliest infectious diseases, with an estimated 10.0 million new cases and 1.6 million deaths in 2017. The World Health Organization (WHO) has set the goal of eliminating TB as a public health problem, aiming to achieve 90% and 95% reductions in the TB incidence and number of TB deaths by 2035. Latent tuberculosis infection (LTBI), a status of persistent immune response to stimulation by Mycobacterium tuberculosis antigens without clinically manifest active TB, has a 10% risk of progressing to active TB and has thus emerged as a critical target for improving TB control and elimination.

The effectiveness of LTBI programmes has long been limited. In 1999, real-world data obtained from an inner-city population in Atlanta, Georgia in the United States revealed that only 27% of subjects receiving isoniazid (INH) preventive therapy completed their treatment. A 2016 meta-analysis including 748,572 subjects in 58 studies also found poor completion of LTBI programmes, with a 60% treatment completion rate. With the introduction of rifapentine (RPT), a rifamycin with much longer half-life than rifampin, the duration of a modern preventive regimen termed 3HP comprising RPT and INH could be shortened to 12 doses administered weekly, with the completion rate approaching 90%. However, 3.8% of those receiving 3HP experience systemic drug reactions (SDRs). The risks of severe adverse event (AE) and SDRs are even higher among subjects >35 years old.

To date, little has been discovered regarding the risk factors or predictors of SDRs due to 3HP therapy. In a pharmacokinetics study of once-weekly RPT treatment in 35 TB patients during continuation phase therapy, serious AEs were not linked with a higher area under the plasma concentration-time curve (AUC0~∞) of RPT. Furthermore, no studies have reported on plasma INH levels after once-weekly INH treatment or the association between plasma INH level and AE development. Under the support of the Taiwan Centers for Disease Control (TCDC), a prospective multicenter observational study was conducted in Taiwan since 2016 to investigate the correlation between SDRs and plasma concentrations of INH, RPT and their major metabolites - acetyl-isoniazid (AcINH) and desacetyl-rifapentine (DeAcRPT). Preliminary results from 129 LTBI cases showed that those with SDRs and those without SDRs had similar plasma concentrations of the 4 compounds at either post-dose 6 or 24 hours (C6 or C24), except that the C24 plasma INH concentration was significantly higher in the SDRs group. Furthermore, generalised estimating equation (GEE) model revealed that C24 plasma INH level was associated with a higher risk of SDR development (OR [95% CI]: 1.61 [1.15-2.25], p = 0.006). By contrast, C24 plasma RPT level was not associated with a higher risk of SDR development (OR [95% CI]: 1.01 [1.00-1.02], p = 0.218).

The 3HP regimen is among the four regimens for LTBI that is recommended by the WHO and is also probably the most promising regimen because of its convenience, with only 12 doses requried. With its effectiveness well established, the major remaining concern regarding 3HP may be its AEs. Studies have estimated that 4.9% to 9.1% of those in close contact with patients with open TB and who received 3HP failed to complete the regimen because of the side effects.8,10 While on the 3HP regimen, SDRs have generally been linked with RPT, which has a well-known side effect: flu-like syndrome. Additionally, RPT is a newer agent, making it a possible contributor to SDRs given that a higher SDR rate was observed compared with other INH-containing regimens. Some scholars, however, have argued against this point. First, one study using the 3HP regimen demonstrated that rechallenge with RPT did not necessarily lead to SDRs. In the same study, rifapentine was better tolerated than isoniazid upon rechallenge. In another study involving 1200 mg of RPT once weekly as continuation therapy for active TB, no SDRs were linked with RPT. Finally, in a study of 162 pulmonary TB patients receiving RPT with a dosage of more than 15mg/kg daily, no patients developed SDRs. In literature review, we discovered that among reports describing an association between RPT and flu-like symptoms, RPT was commonly coadministered with INH. Furthermore, in cases describing an association between INH and flu-like symptoms, the associations were all proven with rechallenge.

Although a less well-known effect than that of RPT, INH can also lead to flu-like syndrome. Of the patients with active TB who were receiving INH, usually with a dose of 300 mg/day, 1%-9.8% developed flu-like syndrome. Case reports describing the association between INH and flu-like syndrome have also been published. In the 3HP regimen, INH dosage is 900 mg/week, and no data exist regarding the proportion of cases developing SDRs under a single INH dosage higher than this.

Some hypotheses could possibly explain the association between the high INH dose and SDRs during 3HP therapy. First, since INH could bind to key enzymes in cytokine pathways such as peroxidase, a high plasma level of INH may activate pathways which are not activated under usual dose of INH due to low binding affinity. Second, the high plasma INH level may interfere with or interact with rifapentine metabolite, resulting in SDRs. Rifapentine, however, did not affect INH pharmacokinetics. Interestingly, a study investigating drug-drug interactions between dolutegravir and once weekly RPT plus INH also revealed a higher INH AUC among those who develop toxicities and a higher INH level among two cases experiencing severe flu-like syndrome. In summary, our preliminary results and recent publications support the association between INH and SDR development because INH drug level, rather than RPT drug level, was discovered to be associated with SDR development, and the short duration and rapid resolution of symptoms in some cases may indicate that a rapidly metabolised drug was the causative agent.

Because rather high doses of INH and RPT are used in 3HP regimen and safety remains a big concern in preventive therapy and program roll-out, a new regimen, consisting of daily INH 300 mg and RPT 600 mg (450 mg if body weight <45.0 kg) for one month was compared with 9H in a large international, open-label RCT enrolling 3000 people living with HIV, so called the BRIEF TB trial. During follow-up, the incidence of active TB was 0.65 vs. 0.67 per 100 person-years in the 1HP and 9H groups, respectively, showing non-inferiority of the ultra-short course of preventive therapy. However, the incidence rate of targeted safety events (liver, gastrointestinal, neurologic, skin or hypersensitivity) was lower with the 1HP regimen (2.9% [2.2 - 3.9%]) than with 9H regimen (4.7% [3.6 - 6.0%], p = 0.016). Treatment completion rates were significantly higher among people taking 1HP (97 vs. 91%, p < 0.01). Because in the PREVENT TB trial the 3HP group had a significantly higher risk of adverse events than the 9H group, the preliminary results of the BRIEF TB trial suggest that by daily use of a relative small dose for both INH and RPT, the 1HP regimen, can be more tolerable than 3HP regimen.

In summary, there remains so many unknowns in rifapentine-based preventive therapy. Further study is necessary to consolidate the finding that INH may play a role in the development of SDRs during 3HP therapy, as well as to evaluate the completion rate and safety profile of 1HP therapy. Therefore, we conduct this prospective multicenter study to investigate whether risk of SDRs under 1HP is lower than that under 3HP.

Research Hypothesis: 1HP has a lower incidence rate of SDRs than 3HP

Objectives:

1. To compare the risk of SDRs in 1HP treatment and in 3HP treatment
2. To explore side effect profile of 1HP

ELIGIBILITY:
Inclusion Criteria:

* aged ≥12 years
* close contact (defined as unprotected exposure of ≥8 hours in a single day or a cumulative duration of ≥40 hours, as per the national policy of Taiwan) with patients diagnosed with acid-fast smear (AFS)-positive pulmonary TB
* diagnosed with LTBI using either a tuberculin skin test (TST) or QuantiFERON-TB Gold in-tube assay (QFT; Cellestis/Qiagen, Carnegie, Australia)

Exclusion Criteria:

* suspected to have active pulmonary TB because of their clinical symptoms or chest radiography findings
* concurrently using drugs with severe drug-drug interactions
* allergic to INH, rifampin, or RPT
* a life expectancy <3 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
number of participants with systemic drug reactions | within 3 months after starting preventive therapy
  AEs that met either of the following: (1) hypotension (systolic blood pressure <90 mm Hg), urticaria, angioedema, acute bronchospasm, or conjunctivitis; and (2) >4 of the following symptoms occurring concurrently (>1 of which had to be grade 2 or higher): weakness, fatigue, nausea, vomiting, headache, fever, aches, sweats, dizziness, shortness of breath, flushing, or chills.

SECONDARY OUTCOMES:
number of participants with any flu-like symptoms | within 3 months after starting preventive therapy
  flu-like symptoms including weakness, fatigue, nausea, vomiting, headache, fever, aches, sweats, dizziness, shortness of breath, flushing, or chills
number of participants with hepatotoxicity | within 3 months after starting preventive therapy
  hepatotoxicity, defined as a 5-fold or greater increase in the AST/ALT level, 3-fold or greater increase with clinical symptoms, or total bilirubin level > 3 mg/dL
Treatment completion rate | within 3 months after starting preventive therapy
  number of participants completing preventive therapy in each arm
Plasma level of isoniazid, rifapentine, acetyl-isoniazid, and Desacetyl-rifapentine | within 3 months after starting preventive therapy
  to investigate whether the occurrence of SDRs is associated with plasma level of isoniazid, rifapentine, acetyl-isoniazid, and desacetyl-rifapentine
Characteristics associated with the development of systemic drug reactions | within 3 months after starting preventive therapy
  to identify the characteristics associated with developing systemic drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Jann-Yuan Wang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang HL, Lee MR, Lee CH, Cheng MH, Lu PL, Sheu CC, Wang JY, Chong IW, Yang JM. One-month daily and three-month weekly rifapentine plus isoniazid are comparable in completion rate and safety for latent tuberculosis infection in non-HIV Population: a randomized controlled trial. Clin Microbiol Infect. 2024 Nov;30(11):1410-1417. doi: 10.1016/j.cmi.2024.06.024. Epub 2024 Jul 10. PMID 38996972